CLINICAL TRIAL: NCT03864614
Title: A Phase 3, Open-Label, 1-Year Study of the Safety, Tolerability, and Need for Re-Treatment With SAGE-217 in Adult Subjects With Major Depressive Disorder
Brief Title: A Study to Evaluate SAGE-217 in Adult Participants With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 217-MDD-303
Record Dates: First submitted 2019-02-05; First posted 2019-03-06 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — zuranolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SAGE-217 (Experimental)
  Interventions: Drug: SAGE-217

INTERVENTIONS:
Drug: SAGE-217 — SAGE-217

SUMMARY:
This is a Phase 3, open-label, 1-year study of the safety, tolerability, and need for re-treatment with SAGE-217 in adult participants with MDD.

DETAILED DESCRIPTION:
This study was previously posted by Sage Therapeutics. In July 2024, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has a diagnosis of MDD as diagnosed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Clinical Trial Version (SCID-5-CT), with symptoms that have been present for at least a 4-week period.
2. Participant is in good physical health and has no clinically significant findings, as determined by the Investigator, on physical examination, 12-lead electrocardiogram (ECG), or clinical laboratory tests.
3. Participant has a Montgomery-Åsberg Depression Rating Scale (MADRS) total score of ≥28 and a HAM-D total score of ≥20 at Screening and Day 1 (prior to dosing).

Exclusion Criteria:

1. Participant has attempted suicide associated with the current episode of MDD.
2. Participant has a medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder.
3. Participant has had vagus nerve stimulation, electroconvulsive therapy, or has taken ketamine (including esketamine) within the current major depressive episode.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1515 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- United States (47):
  - Sage Investigational Site, Dothan, Alabama
  - Sage Investigational Site, Phoenix, Arizona
  - Sage Investigational Site, Anaheim, California
  - Sage Investigational Site, Costa Mesa, California
  - Sage Investigational Site, Glendale, California
  - Sage Investigational Site, Irvine, California
  - Sage Investigational Site, Los Alamitos, California
  - Sage Investigational Site, Oceanside, California
  - Sage Investigational Site, Orange, California
  - Sage Investigational Site, Riverside, California
  - Sage Investigational Site, San Diego, California
  - Sage Investigational Site, Temecula, California
  - Sage Investigational Site, Colorado Springs, Colorado
  - Sage Investigational Site, Cromwell, Connecticut
  - Sage Investigational Site, Norwich, Connecticut
  - Sage Investigational Site, Coral Springs, Florida
  - Sage Investigational Site, Jacksonville, Florida
  - Sage Investigational Site, Miami, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Pensacola, Florida
  - Sage Investigational Site, Alpharetta, Georgia
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Marietta, Georgia
  - Sage Investigational Site, Savannah, Georgia
  - Sage Investigational Site, Chicago, Illinois
  - Sage Investigational Site, Watertown, Massachusetts
  - Sage Investigational Site, Ann Arbor, Michigan
  - Sage Investigational Site, Saint Charles, Missouri
  - Sage Investigational Site, Lincoln, Nebraska
  - Sage Investigational Site, Cherry Hill, New Jersey
  - Sage Investigational site, Marlton, New Jersey
  - Sage Investigational Site, Princeton, New Jersey
  - Sage Investigational Site, Albuquerque, New Mexico
  - Sage Investigational Site, Brooklyn, New York
  - Sage Investigational Site, Mount Kisco, New York
  - Sage Investigational Site, Beachwood, Ohio
  - Sage Investigational Site, Cincinnati, Ohio
  - Sage Investigational site, Cincinnati, Ohio
  - Sage Investigational Site, North Canton, Ohio
  - Sage Investigational Site, Oklahoma City, Oklahoma
  - Sage Investigational Site, Plymouth Meeting, Pennsylvania
  - Sage Investigational Site, Austin, Texas
  - Sage Investigational Site, Dallas, Texas
  - Sage Investigational Site, Houston, Texas
  - Sage Investigational Site, Newport, Texas
  - Sage Investigational Site, Wichita Falls, Texas
  - Sage Investigational Site, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Cutler AJ, Mattingly GW, Kornstein SG, Aaronson ST, Lasser R, Zhang H, Rana N, Brown C, Levin S, Miller C, Kotecha M, Forrestal F, Doherty J. Long-Term Safety and Efficacy of Initial and Repeat Treatment Courses With Zuranolone in Adult Patients With Major Depressive Disorder: Interim Results From the Open-Label, Phase 3 SHORELINE Study. J Clin Psychiatry. 2023 Dec 27;85(1):23m14845. doi: 10.4088/JCP.23m14845. PMID 38153320

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 38 study sites in Part A and 52 study sites in Part B in the United States.
Pre-assignment Details: Participants with Major Depressive Disorder (MDD) were enrolled in this study. This study was conducted in 2 parts, Part A enrolled de novo MDD participants and Part B enrolled MDD participants from the parent study 217- MDD-305 (NCT04476030). Data for Part B was collected and reported in a single arm for each participant who signed informed consent to enroll into this study to be treated with SAGE-217 if and when eligible to be treated.
Groups:
- Part A: Sage-217 High-dose Cohort: Participants received SAGE-217, 50 milligrams (mg), orally, once daily from Day 1 through 14 followed by 14-day follow-up period. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. After the treatment period participants who had a response (a ≥50% reduction from baseline in Hamilton Rating Scale for Depression [HAMD]-17 total score by Day 15) entered a 48-week observational period. During the 48-week observational period, HAMD-17 responders returned to the site every 8 weeks for clinical assessments. Participants were assessed remotely every 14 days via the participant reported 9-item Patient Health Questionnaire (PHQ-9); participants with PHQ-9 score ≥10 returned to the site to be assessed by the clinician administered HAMD-17. If the HAMD-17 total score was ≥20 and 56 days had elapsed since the last dose of the investigational product (IP), the participant began a 14-day SAGE-217 treatment period, which was followed by a 14-day follow-up period
- Part A: Sage-217 Low-dose Cohort: Participants received SAGE-217, 30 mg, orally, once daily from Day 1 through 14 followed by 14-day follow-up period. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. After the treatment period participants who had a response (a ≥50% reduction from baseline in HAMD-17 total score by Day 15) or remission entered a 48-week observational period. During the 48-week observational period, HAMD-17 responders returned to the site every 8 weeks for clinical assessments. Participants were assessed remotely every 14 days via the participant reported 9-item PHQ-9; participants with PHQ-9 score ≥10 returned to the site to be assessed by the clinician administered HAMD-17. If the HAMD-17 total score was ≥20 and 56 days had elapsed since the last dose of the IP, the participant began a 14-day SAGE-217 treatment period, which was followed by a 14-day follow-up period.
- Part A: Sage-217 Dose-switch Cohort: Participants received SAGE-217, 30 mg, orally, once daily in treatment Cycle 1 Day 1 through Day 14 followed by 14-day follow-up period and switched to 50 mg orally, once daily in a subsequent treatment cycle. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. After the treatment period participants who had a response (a ≥50% reduction from baseline in HAMD-17 total score by Day 15) or remission entered a 48-week observational period. During the 48-week observational period, HAMD-17 responders returned to the site every 8 weeks for clinical assessments. Participants were assessed remotely every 14 days via the participant reported 9-item PHQ-9; participants with PHQ-9 score ≥10 returned to the site to be assessed by the clinician administered HAMD-17. If the HAMD-17 total score was ≥20 and 56 days had elapsed since the last dose of the IP, the participant began a 14-day SAGE-217 treatment period, which was followed by a 14-day follow-up period
- Part B: Sage-217: Participants who were eligible to enter the current study from parent study 217-MDD-305 entered the 46-week observational period. Participants were followed with remote assessment of the participant-reported PHQ-9 every 2 weeks; if the PHQ-9 score was ≥10, the participant returned to the site approximately 1 week later and was assessed for the clinician administered HAMD-17. If the HAMD-17 total score was ≥20 and 56 days had elapsed since the last dose of IP, the participant began a 14-day SAGE-217 treatment period, which was followed by a 14-day follow-up period. Participants received SAGE-217 50 mg or 40 mg at the discretion of the investigator, orally, once daily for 14 days followed by 14-day follow-up period. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle.
Period: Overall Study
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort | Part B: Sage-217
Started | 513 | 645 | 80 | 277
Dosed With SAGE-217 Within This Study | 513 | 645 | 80 | 118
Completed | 213 | 236 | 76 | 69
Not Completed | 300 | 409 | 4 | 208
Not completed — Participant Did Not Meet 50% Reduction in HAMD-17 | 116 | 173 | 0 | 0
Not completed — Withdrawal by Subject | 72 | 100 | 1 | 21
Not completed — Lost to Follow-up | 45 | 54 | 0 | 9
Not completed — Adverse Event | 42 | 30 | 1 | 9
Not completed — Protocol Deviation | 6 | 26 | 0 | 1
Not completed — Physician Decision | 7 | 10 | 1 | 5
Not completed — Non-compliance With Investigational Drug | 4 | 4 | 0 | 0
Not completed — Sponsor Decision | 1 | 2 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Other | 7 | 9 | 1 | 4
Not completed — Enrolled but did not receive SAGE-217 | 0 | 0 | 0 | 159

BASELINE CHARACTERISTICS:
Population: For Part A: Safety Set included all participants who were administered SAGE-217. For Part B: Safety Set included participants who signed the informed consent form (ICF) for MDD-303B and had at least 1 dosing of SAGE-217 in the parent study or within MDD-303B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort | Part B: Sage-217 | Total
Number analyzed (Participants) | 513 | 645 | 80 | 190 | 1428
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (15.01) | 44.7 (14.31) | 47.5 (12.71) | 38.9 (12.39) | 43.7 (14.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 331 | 423 | 66 | 127 | 947
  Male | 182 | 222 | 14 | 63 | 481
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 111 | 139 | 37 | 40 | 327
  Not Hispanic or Latino | 402 | 506 | 43 | 150 | 1101
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 1 | 0 | 0 | 7
  Asian | 18 | 22 | 1 | 5 | 46
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 2
  Black or African American | 45 | 108 | 7 | 31 | 191
  White | 432 | 499 | 72 | 153 | 1156
  More than one race | 7 | 11 | 0 | 0 | 18
  Unknown or Not Reported | 4 | 3 | 0 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 513 | 645 | 80 | 190 | 1428

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. For Part A, a TEAE was defined as an AE with onset after the first dose of SAGE-217.
Time Frame: Up to 52 Weeks
Population: Safety Set included all participants who were administered SAGE-217.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Sage-217 High-dose Cohort: Participants received SAGE-217, 50 milligrams (mg), orally, once daily from Day 1 through 14 followed by 14-day follow-up period. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. After the treatment period participants who had a response (a ≥50% reduction from baseline in Hamilton Rating Scale for Depression [HAMD]-17 total score by Day 15) entered a 48-week observational period. During the 48-week observational period, HAMD-17 responders returned to the site every 8 weeks for clinical assessments. Participants were assessed remotely every 14 days via the participant reported 9-item Patient Health Questionnaire (PHQ-9); participants with PHQ-9 score ≥10 returned to the site to be assessed by the clinician administered HAMD-17. If the HAMD-17 total score was ≥20 and 56 days had elapsed since the last dose of the IP, the participant began a 14-day SAGE-217 treatment period, which was followed by a 14-day follow-up period.
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort
Number analyzed (Participants) | 513 | 645 | 80
Participants | 374 | 437 | 57

2. Primary Outcome: Part B: Number of Participants With TEAEs
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. For Part B, a TEAE was defined as an AE with onset on or after the first dose of SAGE-217 in MDD-303B for the participants who received placebo + ADT in parent study, or an AE with onset on or after the ICF signoff in MDD-303B for the participants who received SAGE-217 + ADT in parent study.
Time Frame: Up to 46 Weeks
Population: Study-specific Safety Set included all participants who signed the ICF for 217-MDD-303B and had at least 1 dosing of SAGE-217 within 217-MDD-303B. Data for Part B was collected and reported in a single arm for each participant who started treatment as specified.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Sage-217
Number analyzed (Participants) | 118
Participants | 87

3. Primary Outcome: Part A: Number of Participants With Suicidal Ideation (SI) or Suicidal Behavior (SB) as Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS scale consisted of a baseline evaluation that assessed lifetime experience as well as past 24-month experience of participants for SI and SB and a postbaseline evaluation that focused on suicidality since last study visit. C-SSRS included "yes" or "no"' responses for assessment of SI and SB as well as numeric ratings for severity of ideation, if present. The C-SSRS SI items included: 1. wish to be dead, 2. non-specific active suicidal thoughts, 3. active SI with any methods, 4. active SI with some intent, and 5. active SI with a specific plan (5 being the most severe). C-SSRS SB items included 1. preparatory acts or behavior, 2. aborted attempt, 3. interrupted attempt, 4. actual attempt (non-fatal), and 5. completed suicide (5 being worst). Participants with at least one SI question answered Yes or at least one SB question answered Yes post-baseline for the specific period is counted under SI or SB respectively.
Time Frame: Baseline up to 52 Weeks (Study Period 1-5)
Population: Safety Set included all participants who were administered SAGE-217. For Baseline: Number analyzed is participants of safety set who received SAGE-217 in corresponding study period; For Post-baseline: Number analyzed is participants with data available for analysis at a specific timepoint. A study period is a treatment cycle (treatment period+14-day follow-up) plus the observational period (until next treatment cycle or end of study, whichever is earlier) immediately following it.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort
Number analyzed (Participants) | 513 | 645 | 80
Participants
  Study Period 1: SI: Baseline | 262 | 264 | 29
  Study Period 1: SI: Post-baseline: number analyzed (Participants) | 505 | 642 | 80
  Study Period 1: SI: Post-baseline | 128 | 141 | 14
  Study Period 1: SB: Baseline: number analyzed (Participants) | 513 | 642 | 80
  Study Period 1: SB: Baseline | 6 | 8 | 0
  Study Period 1: SB: Post-baseline: number analyzed (Participants) | 505 | 645 | 80
  Study Period 1: SB: Post-baseline | 3 | 1 | 0
  Study Period 2: SI: Baseline: number analyzed (Participants) | 154 | 206 | 80
  Study Period 2: SI: Baseline | 52 | 57 | 16
  Study Period 2: SI: Post-baseline: number analyzed (Participants) | 154 | 204 | 80
  Study Period 2: SI: Post-baseline | 44 | 51 | 10
  Study Period 2: SB: Baseline: number analyzed (Participants) | 154 | 206 | 80
  Study Period 2: SB: Baseline | 1 | 0 | 0
  Study Period 2: SB: Post-baseline: number analyzed (Participants) | 154 | 204 | 80
  Study Period 2: SB: Post-baseline | 0 | 0 | 0
  Study Period 3: SI: Baseline: number analyzed (Participants) | 74 | 86 | 71
  Study Period 3: SI: Baseline | 16 | 23 | 12
  Study Period 3: SI: Post-baseline: number analyzed (Participants) | 73 | 86 | 71
  Study Period 3: SI: Post-baseline | 17 | 22 | 11
  Study Period 3: SB: Baseline: number analyzed (Participants) | 74 | 86 | 71
  Study Period 3: SB: Baseline | 0 | 0 | 0
  Study Period 3: SB: Post-baseline: number analyzed (Participants) | 73 | 86 | 71
  Study Period 3: SB: Post-baseline | 0 | 0 | 0
  Study Period 4: SI: Baseline: number analyzed (Participants) | 34 | 43 | 53
  Study Period 4: SI: Baseline | 11 | 8 | 10
  Study Period 4: SI: Post-baseline: number analyzed (Participants) | 34 | 43 | 53
  Study Period 4: SI: Post-baseline | 10 | 9 | 9
  Study Period 4: SB: Baseline: number analyzed (Participants) | 34 | 43 | 53
  Study Period 4: SB: Baseline | 0 | 0 | 0
  Study Period 4: SB: Post-baseline: number analyzed (Participants) | 34 | 43 | 53
  Study Period 4: SB: Post-baseline | 1 | 0 | 0
  Study Period 5: SI: Baseline: number analyzed (Participants) | 12 | 20 | 23
  Study Period 5: SI: Baseline | 3 | 1 | 1
  Study Period 5: SI: Post-baseline: number analyzed (Participants) | 12 | 20 | 23
  Study Period 5: SI: Post-baseline | 6 | 3 | 2
  Study Period 5: SB: Baseline: number analyzed (Participants) | 12 | 20 | 23
  Study Period 5: SB: Baseline | 0 | 0 | 0
  Study Period 5: SB: Post-baseline: number analyzed (Participants) | 12 | 20 | 23
  Study Period 5: SB: Post-baseline | 0 | 0 | 0

4. Primary Outcome: Part B: Number of Participants With Suicidal Ideation (SI) and Suicidal Behavior (SB) as Assessed by the C-SSRS
Description: C-SSRS scale consisted of a baseline evaluation that assessed lifetime experience as well as past 24-month experience of participants for SI and SB and a postbaseline (PB) evaluation that focused on suicidality since last study visit. C-SSRS included "yes" or "no"' responses for assessment of SI and SB as well as numeric ratings for severity of ideation, if present. The C-SSRS SI items included: 1. wish to be dead, 2. non-specific active suicidal thoughts, 3. active SI with any methods, 4. active SI with some intent, and 5. active SI with a specific plan (5 being the most severe). C-SSRS SB items included 1. preparatory acts or behavior, 2. aborted attempt, 3. interrupted attempt, 4. actual attempt (non-fatal), and 5. completed suicide (5 being worst). Participants with at least one SI question answered Yes or at least one SB question answered Yes post-baseline for the specific period is counted under SI or SB respectively.
Time Frame: Baseline up to 46 Weeks (Study Period 1-5)
Population: Period-Specific Safety Set included all participants who signed ICF for 217-MDD-303B and were dosed in respective Study Period. A Study Period is a treatment cycle followed by the immediate observation period until the first dose of the subsequent treatment cycle. Data for Part B was collected and reported in a single arm for each participant who started treatment as specified.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Sage-217 All Participants: Participants who were eligible to enter the current study from parent study 217-MDD-305 entered the 46-week observational period. Participants were followed with remote assessment of the participant-reported PHQ-9 every 2 weeks; if the PHQ-9 score was ≥10, the participant returned to the site approximately 1 week later and was assessed for the clinician administered HAMD-17. If the HAMD-17 total score was ≥20 and 56 days had elapsed since the last dose of IP, the participant began a 14-day SAGE-217 treatment period, which was followed by a 14-day follow-up period. Participants received SAGE-217 50 mg or 40 mg at the discretion of the investigator, orally, once daily for 14 days followed by 14-day follow-up period. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle.
Arm/Group | Part B: Sage-217 All Participants
Number analyzed (Participants) | 118
Participants
  Study Period 1: SI: Baseline: number analyzed (Participants) | 57
  Study Period 1: SI: Baseline | 17
  Study Period 1: SI: Post-baseline: number analyzed (Participants) | 57
  Study Period 1: SI: Post-baseline | 16
  Study Period 1: SB: Baseline: number analyzed (Participants) | 57
  Study Period 1: SB: Baseline | 0
  Study Period 1: SB: Post-baseline: number analyzed (Participants) | 57
  Study Period 1: SB: Post-baseline | 1
  Study Period 2: SI: Baseline: number analyzed (Participants) | 87
  Study Period 2: SI: Baseline | 19
  Study Period 2: SI: Post-baseline: number analyzed (Participants) | 87
  Study Period 2: SI: Post-baseline | 24
  Study Period 2: SB: Baseline: number analyzed (Participants) | 87
  Study Period 2: SB: Baseline | 0
  Study Period 2: SB: Post-baseline: number analyzed (Participants) | 87
  Study Period 2: SB: Post-baseline | 0
  Study Period 3: SI: Baseline: number analyzed (Participants) | 44
  Study Period 3: SI: Baseline | 9
  Study Period 3: SI: Post-baseline: number analyzed (Participants) | 44
  Study Period 3: SI: Post-baseline | 9
  Study Period 3: SB: Baseline: number analyzed (Participants) | 44
  Study Period 3: SB: Baseline | 0
  Study Period 3: SB: Post-baseline: number analyzed (Participants) | 44
  Study Period 3: SB: Post-baseline | 0
  Study Period 4: SI: Baseline: number analyzed (Participants) | 20
  Study Period 4: SI: Baseline | 5
  Study Period 4: SI: Post-baseline: number analyzed (Participants) | 20
  Study Period 4: SI: Post-baseline | 6
  Study Period 4: SB: Baseline: number analyzed (Participants) | 20
  Study Period 4: SB: Baseline | 0
  Study Period 4: SB: Post-baseline: number analyzed (Participants) | 20
  Study Period 4: SB: Post-baseline | 0
  Study Period 5: SI: Baseline: number analyzed (Participants) | 5
  Study Period 5: SI: Baseline | 1
  Study Period 5: SI: Post-baseline: number analyzed (Participants) | 5
  Study Period 5: SI: Post-baseline | 1
  Study Period 5: SB: Baseline: number analyzed (Participants) | 5
  Study Period 5: SB: Baseline | 0
  Study Period 5: SB: Post-baseline: number analyzed (Participants) | 5
  Study Period 5: SB: Post-baseline | 0

5. Secondary Outcome: Parts A and B: Time to First Repeat Treatment With SAGE-217
Description: For Part A, the first day of the first repeat treatment is Treatment Cycle 2 Day 1. For Part B, participants who had "placebo + ADT" in the parent study (217-MDD-305), the first repeat treatment of SAGE-217 was the second treatment within MDD-303B. Participants who had SAGE-217 + ADT in the parent study (217-MDD-305), the first repeat treatment of SAGE-217 was the first treatment within MDD-303B. For Part A, as prespecified, data for this outcome measure was collected for Sage-217 High-dose Cohort and Sage-217 30 mg Cohort (Low Dose + Dose Switch). For Part B, data for this outcome measure is presented as per the designated arms in the parent study (217-MDD-305).
  Analysis used Kaplan-Meier estimates where the participants with no repeat treatment were censored.
Time Frame: Up to 52 Weeks
Population: For Part A: FAS included all participants in the Safety Set who had HAMD-17 (change from baseline >=50%) response at Treatment Cycle 1 Day 15 and the discontinuation from study date, if it existed, was after the end of Treatment Cycle 1. For Part B: Safety Set included all participants who received a dose of SAGE-217 either in the parent study 217-MDD-305 or within this protocol 217-MDD-303B.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Part A: Sage-217 30 mg Cohort (Low Dose + Dose Switch): Participants from low-dose cohort (who received 30 mg as first and last dose) and dose-switch cohort (who received 30 mg as their first dose) were included in the 30 mg cohort arm.
- Part B: Placebo + ADT: Participants in the parent study (217-MDD-305) received SAGE-217-matching placebo capsules, orally, once daily along with an assigned anti-depressant therapy (ADT). Participants who were eligible to enter the current study from parent study 217-MDD-305 entered the 46-week observational period. Participants were followed with remote assessment of the participant-reported PHQ-9 every 2 weeks; if the PHQ-9 score was ≥10, the participant returned to the site approximately 1 week later and was assessed for the clinician administered HAMD-17. If the HAMD-17 total score was ≥20 and 56 days had elapsed since the last dose of IP, the participant began a 14-day SAGE-217 treatment period, which was followed by a 14-day follow-up period. Participants received SAGE-217 50 mg or 40 mg at the discretion of the investigator, orally, once daily for 14 days followed by 14-day follow-up period. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle.
- Part B: SAGE-217 + ADT: Participants in the parent study (217-MDD-305) received SAGE-217 capsules, orally, once daily along with an assigned ADT. Participants who were eligible to enter the current study from parent study 217-MDD-305 entered the 46-week observational period. Participants were followed with remote assessment of the participant-reported PHQ-9 every 2 weeks; if the PHQ-9 score was ≥10, the participant returned to the site approximately 1 week later and was assessed for the clinician administered HAMD-17. If the HAMD-17 total score was ≥20 and 56 days had elapsed since the last dose of IP, the participant began a 14-day SAGE-217 treatment period, which was followed by a 14-day follow-up period. Participants received SAGE-217 50 mg or 40 mg at the discretion of the investigator, orally, once daily for 14 days followed by 14-day follow-up period. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle.
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 30 mg Cohort (Low Dose + Dose Switch) | Part B: Placebo + ADT | Part B: SAGE-217 + ADT
Number analyzed (Participants) | 338 | 489 | 57 | 133
days | 281 [191 to NA] — There was no observed failure time (i.e. time to repeat treatment) for which the upper bound of the confidence interval for the Kaplan-Meier estimate is less than 0.5, hence the upper limit of confidence interval remains not estimable. | 135 [121 to 166] | 79 [64 to NA] — There was no observed failure time (i.e. time to repeat treatment) for which the upper bound of the confidence interval for the Kaplan-Meier estimate is less than 0.5, hence the upper limit of confidence interval remains not estimable. | 233 [121 to NA] — There was no observed failure time (i.e. time to repeat treatment) for which the upper bound of the confidence interval for the Kaplan-Meier estimate is less than 0.5, hence the upper limit of confidence interval remains not estimable.

6. Secondary Outcome: Parts A and B: Number of Participants Who Achieved the Requirements for Repeat Treatment for SAGE-217
Description: Participants who continued in the study beyond 56 days from the last study drug dose (in parent study for Part B) and had a HAMD-17 total score ≥20 between the end of first treatment cycle and start of next treatment cycle qualified for repeat treatment for SAGE-217. The 17-item HAM-D was used for measuring severity of depression. It comprised individual ratings of following symptoms scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following symptoms were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score can range from 0 to 52, and higher scores indicated a greater degree of depression. For Part B, data for this outcome measure is presented as per the designated arms in the parent study (217-MDD-305).
Time Frame: Up to 52 Weeks
Population: For Part A: FAS included all participants in the Safety Set who had HAMD-17 response at Treatment Cycle 1 Day 15 and the discontinuation from study date, if it existed, was after the end of Treatment Cycle 1. For Part B: FAS included all participants in the study-specific safety set (dosed at least once within this protocol) who had at least 1 HAMD-17 total score available after the first dose of SAGE-217 within 217-MDD-303B.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Dose-switch Cohort: Participants received SAGE-217, 30 mg, orally, once daily in treatment Cycle 1 Day 1 through Day 14 followed by 14-day follow-up period and switched to 50 mg orally, once daily in a subsequent treatment cycle. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. After the treatment period participants who had a response (a ≥50% reduction from baseline in HAMD-17 total score by Day 15) or remission entered a 48-week observational period. During the 48-week observational period, HAMD-17 responders returned to the site every 8 weeks for clinical assessments. Participants were assessed remotely every 14 days via the participant reported 9-item PHQ-9; participants with PHQ-9 score ≥10 returned to the site to be assessed by the clinician administered HAMD-17. If the HAMD-17 total score was ≥20 and 56 days had elapsed since the last dose of the IP, the participant began a 14-day SAGE-217 treatment period, which was followed by a 14-day follow-up period.
- Part B: Placebo + ADT: Participants in the parent study (217-MDD-305) received SAGE-217-matching placebo capsules, orally, once daily along with an assigned ADT. Participants who were eligible to enter the current study from parent study 217-MDD-305 entered the 46-week observational period. Participants were followed with remote assessment of the participant-reported PHQ-9 every 2 weeks; if the PHQ-9 score was ≥10, the participant returned to the site approximately 1 week later and was assessed for the clinician administered HAMD-17. If the HAMD-17 total score was ≥20 and 56 days had elapsed since the last dose of IP, the participant began a 14-day SAGE-217 treatment period, which was followed by a 14-day follow-up period. Participants received SAGE-217 50 mg or 40 mg at the discretion of the investigator, orally, once daily for 14 days followed by 14-day follow-up period. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle.
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Dose-switch Cohort | Part B: Placebo + ADT | Part B: SAGE-217 + ADT
Number analyzed (Participants) | 338 | 409 | 80 | 57 | 61
Participants | 174 | 224 | 80 | 28 | 61

7. Secondary Outcome: Parts A and B: Number of Repeat Treatment Cycles of SAGE-217 for Each Participant
Description: The response of initial treatment and/or repeat treatment was assessed by HAMD-17. The 17-item HAM-D scale was used for measuring severity of depression. The HAM-D comprised individual ratings of following symptoms scored in range of 0 to 2: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. Following symptoms were scored in range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. total score range=0 to 52, and higher scores indicated greater degree of depression. Participants who had a HAM-D total score >=20 within the protocol were eligible for at least 1 repeat treatment in study. For Part B, data for this outcome measure is presented as per the designated arms in parent study (217-MDD-305). Participants who did not have any re-treatment were included with number of re-treatments equal to 0.
Time Frame: Up to 52 Weeks
Population: For Part A: FAS included all participants in safety set who had HAMD-17 response at Treatment Cycle 1 Day 15 and discontinuation from study date, if it existed, was after end of Treatment Cycle 1. For Part B: FAS included all participants in study-specific safety set (dosed at least once within this protocol) who had at least 1 HAMD-17 total score available after first dose of SAGE-217 within 217-MDD-303B.
Measure: Mean (Standard Deviation); unit: repeat treatment cycles
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort | Part B: Placebo + ADT | Part B: SAGE-217 + ADT
Number analyzed (Participants) | 338 | 409 | 80 | 57 | 61
repeat treatment cycles | 0.8 (1.11) | 0.9 (1.13) | 2.8 (0.97) | 1.6 (0.80) | 1.9 (0.97)

8. Secondary Outcome: Part A: Change From Baseline (CFB) in the HAMD-17 Total Score at Day 15 in Study Period 1
Description: The 17-item HAM-D scale was used for measuring severity of depression. The 17-item HAM-D comprises individual ratings related to the following symptoms: depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early, middle, late), work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. Each item is scored in a range of 0 to 2 or 0 to 4. The total score ranges from 0 to 52 with higher scores indicating a greater degree of depression. A negative change from baseline indicates improvement. A study period is a treatment cycle (treatment period+14-day follow-up) plus the observational period (until next treatment cycle or end of study, whichever is earlier) immediately following it.
Time Frame: Baseline, Day 15 in Study Period 1
Population: The Safety Set was defined as all participants who received SAGE-217. Overall number analyzed is the number of participants with data available for analysis at a specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort
Number analyzed (Participants) | 465 | 607 | 80
score on a scale | -15.3 (6.58) | -14.6 (7.09) | -20.1 (4.61)

9. Secondary Outcome: Part A: Change From Baseline (CFB) in the HAMD-17 Total Score at Day 15 of Each Treatment Cycle
Description: The 17-item HAM-D scale was used for measuring severity of depression. The 17-item HAM-D comprises individual ratings related to the following symptoms: depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early, middle, late), work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. Each item is scored in a range of 0 to 2 or 0 to 4. The total score ranges from 0 to 52 with higher scores indicating a greater degree of depression. A negative change from baseline indicates improvement. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle.
Time Frame: Baseline, Day 15 of treatment cycles 2, 3, 4, and 5
Population: FAS included all participants in the Safety Set who had HAMD-17 response at Treatment Cycle 1 Day 15 and a discontinuation from study date, if it existed, was after the end of Treatment Cycle 1. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at a specific timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort
Number analyzed (Participants) | 150 | 188 | 78
score on a scale
  Treatment cycle 2: CFB at Day 15 | -13.3 (6.36) | -12.3 (6.49) | -15.4 (7.21)
  Treatment cycle 3: CFB at Day 15: number analyzed (Participants) | 69 | 81 | 70
  Treatment cycle 3: CFB at Day 15 | -12.2 (8.06) | -12.5 (6.26) | -15.1 (6.24)
  Treatment cycle 4: CFB at Day 15: number analyzed (Participants) | 34 | 40 | 53
  Treatment cycle 4: CFB at Day 15 | -11.1 (6.42) | -11.7 (7.52) | -15.8 (7.12)
  Treatment cycle 5: CFB at Day 15: number analyzed (Participants) | 12 | 17 | 22
  Treatment cycle 5: CFB at Day 15 | -9.0 (7.17) | -11.6 (6.65) | -17.5 (8.47)

10. Secondary Outcome: Part B: Change From Baseline in the HAMD-17 Total Score at Day 15 of Each Treatment (Initial and/or Repeat Treatment) Cycle
Description: The 17-item HAM-D scale was used to measure the severity of depression. The 17-item HAM-D comprises individual ratings related to the following symptoms: depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early, middle, late), work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. Each item is scored in a range of 0 to 2 or 0 to 4. The total score ranges from 0 to 52 with higher scores indicating a greater degree of depression. A negative change from baseline indicates improvement. Study period is defined as treatment cycle (28 days) followed by immediate observation period (maximum 46 weeks), until the first dose of the subsequent treatment cycle.
Time Frame: Baseline, Day 15 of Study Period 1, 2, 3, 4, and 5
Population: FAS included all participants who signed the ICF for 217-MDD-303B and had at least 1 dosing of SAGE-217 within 217-MDD-303B and had at least 1 HAMD-17 total score available after the first dose of SAGE-217 within 217-MDD-303B. Overall number of participants analyzed is participants in FAS who were dosed in the specific period. Data for this outcome measure was collected and analyzed as per study period.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part B: Study Period 1: Participants who were eligible to enter the current study from parent study 217-MDD-305 entered the 46-week observational period. Participants were followed with remote assessment of the participant-reported PHQ-9 every 2 weeks; if the PHQ-9 score was ≥10, the participant returned to the site approximately 1 week later and was assessed for the clinician administered HAMD-17. If the HAMD-17 total score was ≥20 and 56 days had elapsed since the last dose of IP, the participant began a 14-day SAGE-217 treatment period, which was followed by a 14-day follow-up period. Participants received SAGE-217 50 mg or 40 mg at the discretion of the investigator, orally, once daily for 14 days followed by 14-day follow-up period. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. Study Period 1 included only placebo + ADT participants from the parent study (217-MDD-305).
- Part B: Study Period 2: Participants received SAGE-217 50 mg or 40 mg at the discretion of the investigator, orally, once daily for 14 days followed by 14-day follow-up period. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. After the treatment period participants who had a response (a ≥50% reduction from baseline in HAMD-17 total score by Day 15) or remission entered a 46-week observational period. During the 46-week observational period, HAMD-17 responders returned to the site every 8 weeks for clinical assessments. Participants were assessed remotely every 14 days via the participant reported 9-item PHQ-9; participants with PHQ-9 score ≥10 returned to the site to be assessed by the clinician administered HAMD-17. At Day 70 or later, participants with a HAMD-17 total score ≥20, assessed approximately 1 week from the PHQ-9 score ≥10, were eligible for repeat treatment. Study Period 2 included both placebo + ADT and SAGE 217 + ADT participants from the parent study (217-MDD-305).
- Part B: Study Period 3: Participants received SAGE-217 50 mg or 40 mg at the discretion of the investigator, orally, once daily for 14 days followed by 14-day follow-up period. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. After the treatment period participants who had a response (a ≥50% reduction from baseline in HAMD-17 total score by Day 15) or remission entered a 46-week observational period. During the 46-week observational period, HAMD-17 responders returned to the site every 8 weeks for clinical assessments. Participants were assessed remotely every 14 days via the participant reported 9-item PHQ-9; participants with PHQ-9 score ≥10 returned to the site to be assessed by the clinician administered HAMD-17. At Day 70 or later, participants with a HAMD-17 total score ≥20, assessed approximately 1 week from the PHQ-9 score ≥10, were eligible for repeat treatment. Study Period 3 included both placebo + ADT and SAGE 217 + ADT participants from the parent study (217-MDD-305).
- Part B: Study Period 4: Participants received SAGE-217 50 mg or 40 mg at the discretion of the investigator, orally, once daily for 14 days followed by 14-day follow-up period. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. After the treatment period participants who had a response (a ≥50% reduction from baseline in HAMD-17 total score by Day 15) or remission entered a 46-week observational period. During the 46-week observational period, HAMD-17 responders returned to the site every 8 weeks for clinical assessments. Participants were assessed remotely every 14 days via the participant reported 9-item PHQ-9; participants with PHQ-9 score ≥10 returned to the site to be assessed by the clinician administered HAMD-17. At Day 70 or later, participants with a HAMD-17 total score ≥20, assessed approximately 1 week from the PHQ-9 score ≥10, were eligible for repeat treatment. Study Period 4 included both placebo + ADT and SAGE 217 + ADT participants from the parent study (217-MDD-305).
- Part B: Study Period 5: Participants received SAGE-217 50 mg or 40 mg at the discretion of the investigator, orally, once daily for 14 days followed by 14-day follow-up period. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. After the treatment period participants who had a response (a ≥50% reduction from baseline in HAMD-17 total score by Day 15) or remission entered a 46-week observational period. During the 46-week observational period, HAMD-17 responders returned to the site every 8 weeks for clinical assessments. Participants were assessed remotely every 14 days via the participant reported 9-item PHQ-9; participants with PHQ-9 score ≥10 returned to the site to be assessed by the clinician administered HAMD-17. At Day 70 or later, participants with a HAMD-17 total score ≥20, assessed approximately 1 week from the PHQ-9 score ≥10, were eligible for repeat treatment. Study Period 5 included only SAGE 217 + ADT participants from the parent study (217-MDD-305).
Arm/Group | Part B: Study Period 1 | Part B: Study Period 2 | Part B: Study Period 3 | Part B: Study Period 4 | Part B: Study Period 5
Number analyzed (Participants) | 52 | 85 | 42 | 20 | 5
score on a scale | -10.1 (6.43) | -10.7 (6.49) | -9.6 (7.53) | -9.7 (7.60) | -10.8 (9.26)

11. Secondary Outcome: Part A: Percentage of Participants Who Achieved HAM-D Response During Treatment Cycle 1
Description: HAM-D response was defined as a ≥50% reduction in HAM-D score from baseline, at the end of each 14-day treatment period. The 17-item HAM-D scale was used for measuring severity of depression. The HAM-D comprised individual ratings of the following symptoms scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following symptoms were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score can range from 0 to 52, and higher scores indicated a greater degree of depression. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. Percentage are rounded off.
Time Frame: Day 15 of treatment cycle 1
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort
Number analyzed (Participants) | 513 | 645 | 80
percentage of participants | 67.3 | 65.9 | 100

12. Secondary Outcome: Part A: Percentage of Participants Who Achieved HAM-D Response During Each Study Period
Description: HAM-D response was defined as a ≥50% reduction in HAM-D score from baseline, at the end of each 14-day treatment period. The 17-item HAM-D scale was used for measuring severity of depression. The HAM-D comprised individual ratings of the following symptoms scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following symptoms were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score can range from 0 to 52, and higher scores indicated a greater degree of depression. A study period is a treatment cycle (treatment period+14-day follow-up) plus the observational period (until next treatment cycle or end of study, whichever is earlier) immediately following it. Percentage are rounded off.
Time Frame: Day 15 of Study Period 2, 3, 4, and 5
Population: FAS included all participants in the Safety Set who had HAMD-17 response at Treatment Cycle 1 Day 15 and the discontinuation from study date, if it existed, was after the end of Treatment Cycle 1. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort
Number analyzed (Participants) | 150 | 188 | 78
percentage of participants
  Study Period 2: Day 15 | 65.3 | 62.8 | 67.9
  Study Period 3: Day 15: number analyzed (Participants) | 69 | 81 | 70
  Study Period 3: Day 15 | 58.0 | 59.3 | 68.6
  Study Period 4: Day 15: number analyzed (Participants) | 34 | 40 | 53
  Study Period 4: Day 15 | 38.2 | 55.0 | 75.5
  Study Period 5: Day 15: number analyzed (Participants) | 12 | 17 | 22
  Study Period 5: Day 15 | 25.0 | 58.8 | 81.8

13. Secondary Outcome: Part B: Percentage of Participants Who Achieved HAM-D Response
Description: HAM-D response was defined as a ≥50% reduction in HAM-D score from baseline, at the end of each 14-day treatment period. The 17-item HAM-D scale was used for measuring severity of depression. The HAM-D comprised individual ratings of the following symptoms scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following symptoms were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score can range from 0 to 52, and higher scores indicated a greater degree of depression. A study period is defined as treatment cycle (28 days) followed by immediate observation period (maximum 46 weeks), until the first dose of the subsequent treatment cycle. Percentage are rounded off.
Time Frame: Day 15 of Study Period 1, 2, 3, 4, and 5
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Study Period 1 | Part B: Study Period 2 | Part B: Study Period 3 | Part B: Study Period 4 | Part B: Study Period 5
Number analyzed (Participants) | 52 | 85 | 42 | 20 | 5
percentage of participants | 46.2 | 47.1 | 38.1 | 30.0 | 60.0

14. Secondary Outcome: Part A: Percentage of Participants Who Achieved HAM-D Remission During Treatment Cycle 1
Description: Remission was defined as having a HAM-D total score of ≤7. The 17-item HAM-D scale was used for measuring severity of depression. The HAM-D comprised individual ratings of the following symptoms scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following symptoms were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score can range from 0 to 52, and higher scores indicated a greater degree of depression. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. Percentage are rounded off.
Time Frame: Day 15 of treatment cycle 1
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort
Number analyzed (Participants) | 465 | 607 | 80
percentage of participants | 40.9 | 40.2 | 40.0

15. Secondary Outcome: Part A: Percentage of Participants Who Achieved HAM-D Remission During Each Study Period
Description: Remission was defined as having a HAM-D total score of ≤7. The 17-item HAM-D scale was used for measuring severity of depression. The HAM-D comprised individual ratings of the following symptoms scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following symptoms were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score can range from 0 to 52, and higher scores indicated a greater degree of depression. A study period is a treatment cycle (treatment period+14-day follow-up) plus the observational period (until next treatment cycle or end of study, whichever is earlier) immediately following it. Percentage are rounded off.
Time Frame: Day 15 of Study Periods 2, 3, 4, and 5
Population: FAS included all participants in the Safety Set who had HAMD-17 response at Treatment Cycle 1 Day 15 and the discontinuation from study date, if it existed, was after the end of Treatment Cycle 1. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available at a given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort
Number analyzed (Participants) | 150 | 188 | 78
percentage of participants
  Study Period 2: Day 15 | 38.7 | 31.9 | 37.2
  Study Period 3: Day 15: number analyzed (Participants) | 69 | 81 | 70
  Study Period 3: Day 15 | 34.8 | 29.6 | 32.9
  Study Period 4: Day 15: number analyzed (Participants) | 34 | 40 | 53
  Study Period 4: Day 15 | 23.5 | 32.5 | 43.4
  Study Period 5: Day 15: number analyzed (Participants) | 12 | 17 | 22
  Study Period 5: Day 15 | 16.7 | 29.4 | 63.6

16. Secondary Outcome: Part B: Percentage of Participants Who Achieved HAM-D Remission
Description: Remission was defined as having a HAM-D total score of ≤7. The 17-item HAM-D scale was used for measuring severity of depression. The HAM-D comprised individual ratings of the following symptoms scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following symptoms were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score can range from 0 to 52, and higher scores indicated a greater degree of depression. A Study Period is defined as Treatment Cycle (28 days) followed by the immediate observational period (maximum 46 weeks), until the first dose of the subsequent treatment cycle. Percentage are rounded off.
Time Frame: Day 15 of Study Period 1, 2, 3, 4, and 5
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Study Period 1 | Part B: Study Period 2 | Part B: Study Period 3 | Part B: Study Period 4 | Part B: Study Period 5
Number analyzed (Participants) | 52 | 85 | 42 | 20 | 5
percentage of participants | 19.2 | 29.4 | 26.2 | 20.0 | 40.0

17. Secondary Outcome: Part A: Percentage of Participants Who Achieved Clinical Global Impression - Improvement (CGI-I) Response During Treatment Cycle 1
Description: The CGI scale consists of 3 items. Only the first 2 items are being used in this study. The CGI-I employed a 7-point Likert scale to measure the overall improvement in the participant's condition posttreatment. The Investigator rated the participant's total improvement compared to baseline, whether or not it was due entirely to drug treatment. Response choices included: 0=not assessed, 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse. The CGI-I is only rated at posttreatment assessments. CGI-I response was defined as having a CGI-I score of "very much improved" or "much improved." Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. Percentage are rounded off.
Time Frame: Day 15 of treatment cycle 1
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort
Number analyzed (Participants) | 464 | 608 | 80
percentage of participants | 78.9 | 75.0 | 96.3

18. Secondary Outcome: Part A: Percentage of Participants Who Achieved CGI-I Response During Each Study Period
Description: The CGI scale consists of 3 items. Only the first 2 items are being used in this study. The CGI-I employed a 7-point Likert scale to measure the overall improvement in the participant's condition posttreatment. The Investigator rated the participant's total improvement compared to baseline, whether or not it was due entirely to drug treatment. Response choices included: 0=not assessed, 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse. The CGI-I is only rated at posttreatment assessments. CGI-I response was defined as having a CGI-I score of "very much improved" or "much improved." A study period is a treatment cycle (treatment period+14-day follow-up) plus the observational period (until next treatment cycle or end of study, whichever is earlier) immediately following it. Percentage are rounded off.
Time Frame: Day 15 of Study Periods 2, 3, 4, and 5
Population: FAS included all participants in the Safety Set who had HAMD-17 response at Treatment Cycle 1 Day 15 and the discontinuation from study date, if it existed, was after the end of Treatment Cycle 1. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at specific timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort
Number analyzed (Participants) | 150 | 188 | 78
percentage of participants
  Study Period 2: Day 15 | 76.7 | 75.0 | 79.5
  Study Period 3: Day 15: number analyzed (Participants) | 69 | 82 | 68
  Study Period 3: Day 15 | 65.2 | 73.2 | 80.9
  Study Period 4: Day 15: number analyzed (Participants) | 34 | 40 | 53
  Study Period 4: Day 15 | 52.9 | 60.0 | 84.9
  Study Period 5: Day 15: number analyzed (Participants) | 12 | 16 | 22
  Study Period 5: Day 15 | 33.3 | 68.8 | 90.9

19. Secondary Outcome: Part B: Percentage of Participants Who Achieved CGI-I Response
Description: The CGI scale consists of 3 items. Only the first 2 items are being used in this study. The CGI-I employed a 7-point Likert scale to measure the overall improvement in the participant's condition posttreatment. The Investigator rated the participant's total improvement compared to baseline, whether or not it was due entirely to drug treatment. Response choices included: 0=not assessed, 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse. The CGI-I is only rated at posttreatment assessments. CGI-I response was defined as having a CGI-I score of "very much improved" or "much improved." A Study Period is defined as Treatment Cycle (28 days) followed by the immediate observational period (maximum 46 weeks), until the first dose of the subsequent treatment cycle. Percentage are rounded off.
Time Frame: Day 15 of Study Period 1, 2, 3, 4, and 5
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Study Period 1 | Part B: Study Period 2 | Part B: Study Period 3 | Part B: Study Period 4 | Part B: Study Period 5
Number analyzed (Participants) | 52 | 85 | 42 | 20 | 5
percentage of participants | 53.8 | 63.5 | 64.3 | 55.0 | 60.0

20. Secondary Outcome: Part A: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score During Treatment Cycle 1
Description: The CGI-S uses a 7-point Likert scale to rate the severity of the participant's mental illness at the time of assessment, relative to the clinician's past experience with participants who had the same diagnosis. Considering total clinical experience, a participant was assessed on severity of mental illness at the time of rating as 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=extremely ill. A higher score indicated extreme illness. A negative change from baseline indicated improvement. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle.
Time Frame: Baseline, Day 15 of treatment cycle 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort
Number analyzed (Participants) | 464 | 608 | 80
score on a scale | -2.3 (1.22) | -2.1 (1.25) | -2.4 (1.01)

21. Secondary Outcome: Part A: Change From Baseline in CGI-S Score During Each Treatment Cycle
Description: as for outcome 20
Time Frame: Baseline, Day 15 of treatment cycles 2, 3, 4, and 5
Population: FAS included all participants in the Safety Set who had HAMD-17 response at Treatment Cycle 1 Day 15 and the discontinuation from study date, if it existed, was after the end of Treatment Cycle 1. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at specific timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort
Number analyzed (Participants) | 150 | 188 | 78
score on a scale
  Treatment Cycle 2: CFB at Day 15 | -2.0 (1.15) | -1.9 (1.23) | -2.2 (1.43)
  Treatment Cycle 3: CFB at Day 15: number analyzed (Participants) | 69 | 82 | 68
  Treatment Cycle 3: CFB at Day 15 | -1.8 (1.32) | -1.8 (1.21) | -2.1 (1.35)
  Treatment Cycle 4: CFB at Day 15: number analyzed (Participants) | 34 | 40 | 53
  Treatment Cycle 4: CFB at Day 15 | -1.8 (1.16) | -1.7 (1.33) | -2.4 (1.64)
  Treatment Cycle 5: CFB at Day 15: number analyzed (Participants) | 12 | 16 | 22
  Treatment Cycle 5: CFB at Day 15 | -1.2 (1.27) | -1.9 (1.09) | -2.7 (1.83)

22. Secondary Outcome: Part B: Change From Baseline in CGI-S Score
Description: The CGI-S uses a 7-point Likert scale to rate the severity of the participant's mental illness at the time of assessment, relative to the clinician's past experience with participants who had the same diagnosis. Considering total clinical experience, a participant was assessed on severity of mental illness at the time of rating as 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=extremely ill. A higher score indicated extreme illness. A negative change from baseline indicated improvement. A Study Period is defined as Treatment Cycle (28 days) followed by the immediate observational period (maximum 46 weeks), until the first dose of the subsequent treatment cycle.
Time Frame: Baseline Day 15 of Study Period 1, 2, 3, 4, and 5
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Study Period 1 | Part B: Study Period 2 | Part B: Study Period 3 | Part B: Study Period 4 | Part B: Study Period 5
Number analyzed (Participants) | 52 | 85 | 42 | 20 | 5
score on a scale | -1.5 (1.18) | -1.8 (1.15) | -1.7 (1.26) | -1.4 (1.39) | -1.4 (1.52)

ADVERSE EVENTS:
Time Frame: For Part A: Up to 52 Weeks; For Part B: Up to 46 Weeks
Description: For Part A: Safety Set included all participants who were administered SAGE-217; For Part B: Study-specific Safety Set included all participants who were administered SAGE-217 within 217-MDD-303B. Data for Part B was collected and reported in a single arm for each participant who started treatment as specified.
Groups:
- Part A: Sage-217 High-dose Cohort: Participants received SAGE-217, 50 mg, orally, once daily from Day 1 through 14 followed by 14-day follow-up period. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. After the treatment period participants who had a response (a ≥50% reduction from baseline in HAMD-17 total score by Day 15) or remission entered a 48-week observational period. During the 48-week observational period, HAMD-17 responders returned to the site every 8 weeks for clinical assessments. Participants were assessed remotely every 14 days via the participant reported 9-item PHQ-9; participants with PHQ-9 score ≥10 returned to the site to be assessed by the clinician administered HAMD-17. At Day 70 or later, participants with a HAMD-17 total score ≥20, assessed approximately 1 week from the PHQ-9 score ≥10, were eligible for repeat treatment.
- Part A: Sage-217 Low-dose Cohort: Participants received SAGE-217, 30 mg, orally, once daily from Day 1 through 14 followed by 14-day follow-up period. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. After the treatment period participants who had a response (a ≥50% reduction from baseline in HAMD-17 total score by Day 15) or remission entered a 48-week observational period. During the 48-week observational period, HAMD-17 responders returned to the site every 8 weeks for clinical assessments. Participants were assessed remotely every 14 days via the participant reported 9-item PHQ-9; participants with PHQ-9 score ≥10 returned to the site to be assessed by the clinician administered HAMD-17. At Day 70 or later, participants with a HAMD-17 total score ≥20, assessed approximately 1 week from the PHQ-9 score ≥10, were eligible for repeat treatment.
- Part A: Sage-217 Dose-switch Cohort: Participants received SAGE-217, 30 mg, orally, once daily in treatment Cycle 1 Day 1 through Day 14 followed by 14-day follow-up period and switched to 50 mg orally, once daily in a subsequent treatment cycle. Each 14-day treatment period plus corresponding 14-day follow-up period was considered a treatment cycle. After the treatment period participants who had a response (a ≥50% reduction from baseline in HAMD-17 total score by Day 15) or remission entered a 48-week observational period. During the 48-week observational period, HAMD-17 responders returned to the site every 8 weeks for clinical assessments. Participants were assessed remotely every 14 days via the participant reported 9-item PHQ-9; participants with PHQ-9 score ≥10 returned to the site to be assessed by the clinician administered HAMD-17. At Day 70 or later, participants with a HAMD-17 total score ≥20, assessed approximately 1 week from the PHQ-9 score ≥10, were eligible for repeat treatment.
Arm/Group | Part A: Sage-217 High-dose Cohort | Part A: Sage-217 Low-dose Cohort | Part A: Sage-217 Dose-switch Cohort | Part B: Sage-217 All Participants
All-Cause Mortality (participants affected / at risk) | 0/513 | 1/645 | 0/80 | 0/118
Serious Adverse Events (participants affected / at risk) | 18/513 | 19/645 | 1/80 | 4/118
Other Adverse Events (participants affected / at risk) | 371/513 | 435/645 | 57/80 | 87/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Sage-217 High-dose Cohort (N=513) | Part A: Sage-217 Low-dose Cohort (N=645) | Part A: Sage-217 Dose-switch Cohort (N=80) | Part B: Sage-217 All Participants (N=118)
Suicidal ideation (Psychiatric disorders) | 2 | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 2 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Herpes simplex encephalitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Breast necrosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Sage-217 High-dose Cohort (N=513) | Part A: Sage-217 Low-dose Cohort (N=645) | Part A: Sage-217 Dose-switch Cohort (N=80) | Part B: Sage-217 All Participants (N=118)
Somnolence (Nervous system disorders) | 102 | 76 | 10 | 19
Headache (Nervous system disorders) | 61 | 90 | 13 | 13
Dizziness (Nervous system disorders) | 78 | 47 | 7 | 13
Sedation (Nervous system disorders) | 57 | 29 | 11 | 8
Tremor (Nervous system disorders) | 28 | 9 | 3 | 0
Migraine (Nervous system disorders) | 6 | 6 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 26 | 43 | 11 | 6
Dry mouth (Gastrointestinal disorders) | 22 | 40 | 3 | 0
Nausea (Gastrointestinal disorders) | 28 | 25 | 3 | 9
Dyspepsia (Gastrointestinal disorders) | 5 | 18 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 23 | 52 | 5 | 9
COVID-19 (Infections and infestations) | 44 | 2 | 3 | 9
Insomnia (Psychiatric disorders) | 23 | 31 | 5 | 8
Anxiety (Psychiatric disorders) | 17 | 19 | 4 | 0
Fatigue (General disorders) | 22 | 27 | 8 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 18 | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 14 | 5 | 0
Vertigo (Ear and labyrinth disorders) | 8 | 5 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (3):
  • Study Protocol (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03864614/Prot_000.pdf
  • Statistical Analysis Plan: Part A: Statistical Analysis Plan (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT03864614/SAP_001.pdf
  • Statistical Analysis Plan: Part B: Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT03864614/SAP_002.pdf